CLINICAL TRIAL: NCT01755533
Title: Adaptation Processes in School-Based Substance Abuse Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Ohio State University (Other)
Responsible Party: Principal Investigator, Michael L. Hecht, Distinguished Professor of Communication Arts and Sciences, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DESPR DA021670; R01DA021670 (NIH)
Record Dates: First submitted 2012-12-21; First posted 2012-12-24 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Substance Use
Keywords: adolescent substance use; rural substance use; middle school prevention; implementation processes; implementation quality; adaptation of prevention curricula; dissemination
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rural curriculum (Experimental): Receive rural version of curriculum
  Interventions: Other: Rural curriculum
- Classic curriculum (Experimental): Receive classic version of curriculum
  Interventions: Other: Classic curriculum
- Control (No Intervention): Continue normal prevention activities

INTERVENTIONS:
Other: Rural curriculum — Students in schools randomly assigned to this condition receive the rural version of the curriculum.
  Arms: Rural curriculum
Other: Classic curriculum — Students in schools randomly assigned to this condition receive the classic version of the curriculum.
  Arms: Classic curriculum

SUMMARY:
The goals of this study are to develop a middle school substance use prevention curriculum for underserved rural youth and evaluate its efficacy compared to the existing, multicultural curriculum. In addition, we are studying how the curricula get taught by the teachers.

Hypothesis 1: When compared to students in the control condition, students in the treatment conditions will report less substance use, more conservative norms, less positive expectations about substance use outcomes, and better life and communication skills.

Hypothesis 2: When compared to students in the control condition, students in the researcher adaptation condition will report less substance use, more conservative norms, less positive expectations, and better life and communication skills.

Hypothesis 3: When compared to students in the control condition, students in the teacher adaptation condition will report less substance use, more conservative norms, less positive expectations, and better life and communication skills.

Hypothesis 4: Researcher adaptation will have a greater impact on substance use, norms, and expectations than teacher adaptation.

DETAILED DESCRIPTION:
The goals of the proposed study are to conduct an effectiveness trial of the keepin' it REAL middle school substance use prevention curriculum among a new target audience in rural Pennsylvania and Ohio, describe how teachers adapt the curriculum when they present it, and develop, implement, and evaluate a Pennsylvania/Ohio-version of the curriculum to test whether an evidence-based universal curriculum can be improved by adapting it to local cultures. keepin' it REAL is recognized as a "model program" by SAMHSA's National Registry of Effective programs and is one of the few that are multicultural. The study will evaluate the effectiveness of the original curriculum, grounded in the cultures of the southwest and compare that to a new version, "regrounded" in the rural culture of Pennsylvania and Ohio, while studying how teachers adapt both versions. This proposal responds to NIDA PA-05-118, Drug Abuse Prevention Intervention Research that calls for investigations addressing, "1) the development of novel drug abuse prevention approaches; 2) the efficacy and effectiveness of newly developed and/or modified prevention programs; 3) the processes associated with the selection, adoption, adaptation, implementation, sustainability, and financing of empirically validated interventions." This proposal addresses all three points.

A randomized control trial will be conducted in middle schools to accomplish these goals. First, formative research will be conducted to develop a rural Pennsylvania/Ohio-version of the curriculum. Second, 42 rural schools will be randomly assigned to one of three conditions: teacher adaptation in which the original keepin' it REAL curriculum is implemented; researcher adaptation in which a new Pennsylvania-version of the curriculum is implemented, and a control group. We hypothesized the participation in either form of the curriculum will reduce drug use and that the researcher adaptation will produce better outcomes and less teacher adaptation than the teacher adaptation. A pretest will be administered followed by posttests in 7-9th grades. Adaptation and fidelity will be measured in 3 ways: teachers completing a Program Quality and Adaptation online measure after each lesson, videotaped lessons, and attendance. The major hypothesis tests will be conducted using variants of the general linear model, taking into account the multilevel structure of the data (e.g., multilevel multiple regression), test of a mediation model, and growth modeling.

ELIGIBILITY:
Inclusion Criteria:

* Any student enrolled in treatment or control classes

Exclusion Criteria:

* Students not enrolled in treatment or control classes

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2827 (Actual)
Dates: Start 2008-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in substance use | Between the beginning of 7th grade and the end of 9th grade
  Self report measure

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Hecht, PhD, Principal Investigator — Penn State University
Locations (1):
- Department of Communication Arts & Sciences, Penn State University, University Park, Pennsylvania, United States

REFERENCES:
- [Result] Pettigrew J, Miller-Day M, Krieger J, Hecht ML. Alcohol and Other Drug Resistance Strategies Employed by Rural Adolescents. J Appl Commun Res. 2011;39(2):103-122. doi: 10.1080/00909882.2011.556139. PMID 21552345